CLINICAL TRIAL: NCT07288112
Title: Clinical Study of DOC1021 Dendritic Cell Immunotherapy for Refractory Melanoma
Brief Title: DOC1021 Dendritic Cell Immunotherapy for Refractory Melanoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Diakonos Oncology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC-RM
Record Dates: First submitted 2025-12-03; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Refractory Melanoma
Keywords: Dendritic Cell Vaccine; Immunotherapy; Tumor Vaccine
MeSH Terms: conditions — Melanoma | interventions — Transurethral Resection of Bladder; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: DOC1021 + pIFN (Experimental): DOC1021 administered by injection near active tumor lesion lymph nodes + pIFN
  Interventions: Biological: DOC1021; Procedure: Tumor resection; Drug: pIFN (peginterferon alfa-2a)

INTERVENTIONS:
Biological: DOC1021 — Double-loaded dendritic cell vaccine, loaded with tumor lysate and mRNA using proprietary method
Procedure: Tumor resection — Tumor resection or biopsy
Drug: pIFN (peginterferon alfa-2a) — pIFN 180 mcg subcutaneously every week for 4 total doses

SUMMARY:
The goal of this clinical trial is to learn if DOC1021 + pIFN will be safe and will lead to tumor responses in patients with refractory melanoma. DOC1021 is a dendritic cell immunotherapy derived from a patient's own blood cells and loaded with antigens from the patient's tumor in the form of tumor lysate and mRNA. The goal is to stimulate a T cell immune response that eliminates tumor cells.

The study consists of two components: an initial phase I safety study to confirm safety/tolerability of the treatment regimen, and, subsequently, a single-arm phase II cohort to assess efficacy of the treatment regimen.

All participants will:

* Take filgrastim subcutaneously x 5 doses and subsequently undergo a leukapheresis collection
* Receive two doses of DOC1021 under image guidance 2 weeks apart
* Receive subcutaneous pIFN injections weekly for a total of 4 doses in parallel with the DOC1021 injections
* Undergo an optional image-guided perinodal DOC1021 booster injection approximately 6 months after the first DOC1021 dose along with additional subcutaneous pIFN injections at time of the booster and the subsequent week for a total of 2 pIFN doses
* Visit the clinic regularly to assess quality of life, symptoms, medication use, imaging, bloodwork, and to receive optional treatment with anti-PD1 agents

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and avail-ability for the duration of the study
3. Age 18 years or older
4. Patients diagnosed with unresectable or metastatic melanoma and progressed following ≥1 prior systemic therapy including anti-PD-1 (i.e., refractory to anti-PD-1). Refractory defined as primary or secondary resistance as per SITC guidelines, except that confirmatory scan not required if clinical progression requiring surgery or radiation to relieve symptoms
5. Willing and able to withhold anti-PD-1 treatment from the time of enrollment through ~6 weeks after the first DOC1021 administration
6. One or more lesions available for biopsy or resection to yield at least 50 mg (e.g., 5 core biopsies) and preferably 100 mg of tumor for generating DOC1021 and at least 1 measurable target tumor lesion evaluable after DOC1021 by RECIST version 1.1.
7. Brain metastases allowed if stable after prior treatment
8. Ability to receive filgrastim (e.g. Neupogen), leukapheresis and perinodal injections of DOC1021 near regional nodes + weekly pIFN x 4 weeks.
9. Females of reproductive potential must have a negative serum pregnancy test and agree to use effective contraception (as deter-mined appropriate for the patient by the investigator) during study treatment.
10. Adequate kidney, liver, bone marrow function, and immune function, as follows:

    1. Hemoglobin ≥ 8.0 gm/dL (use of transfusion or other intervention to achieve is acceptable)
    2. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
    3. Platelet count ≥ 75,000/mm3
    4. Calculated creatinine clearance (CrCl) > 30 mL/min using Cockcroft and Gault formula:

    i. For males = (140 - age[years]) x (body weight [kg]) / (72 x serum creatinine [mg/dL]) ii. For females = 0.85 x value from male formula e. Total bilirubin ≤ 1.5 times upper limit of normal (ULN) except in patients with Gilbert's disease for which total bilirubin must be ≤ 3 times ULN f. Aspartate transaminase AST (SGOT) and alanine aminotransferase ALT (SGPT) ≤ 3 times the ULN (or ≤ 5.0 × ULN if liver metastases)
11. Eastern Cooperative Group (ECOG) Performance Score 0 or 1

Exclusion Criteria:

1. Patients who are pregnant or breastfeeding.
2. Known active HIV or hepatitis infection. Patients with HIV that is well-controlled and have undetectable viral titers remain eligible. Patients with history of HCV adequately treated such that RNA viral load is negative also remain eligible.
3. Any severe or uncontrolled medical condition or other condition that could affect participation in this study as determined by the investigator, including but not limited to uncontrolled or severe cardiac dis-ease, systemic autoimmune disorders requiring immunosuppression*, autoimmune hyper/hypothyroidism, untreated viral hepatitis, autoimmune hepatitis (*autoimmune disorders include but are not limited to rheumatoid arthritis, psoriasis and inflammatory bowel disease and immunosuppressive medications include DMARDs like methotrexate, TNF inhibitors, IL-6 receptor blockers, CD80/86 inhibitors, anti-CD20 and JAK inhibitors)
4. Residual immune-related toxicities from prior immunotherapy > Grade 1 severity. However, patients who experienced prior endocrine toxicity are eligible if well-controlled on replacement therapy.
5. Treatment with another investigational drug or other experimental intervention within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: To evaluate the number of dose limiting toxicities reported | From time of first DOC1021 dose administration to 6 weeks later
Phase II: To evaluate the objective response rate (ORR) as the proportion of patients with a confirmed complete response (CR) or partial response (PR) to treatment, as per RECIST 1.1 criteria | 5 years

SECONDARY OUTCOMES:
Overall survival (time in months from the date of study enrollment until death for from any cause) | 5 years
Time in months from the first documentation of complete or partial response to disease progression by RECIST 1.1 criteria or death, whichever occurs first. | 5 years
  Duration of Response (DOR)
Time in months from date of study enrollment to disease progression by RECIST 1.1 criteria or death from any cause | 3 years
  Progression-free survival (PFS)
The proportion of participants with complete response, partial response, or stable disease out of the total eligible and evaluable participants. | 5 years
  Disease control rate (DCR)
Number of participants with adverse events as assessed by CTCAE v5.0 | 3 years
To evaluate the objective response rate (ORR) as the proportion of patients with a confirmed complete response (CR) or partial response (PR) to treatment, as per immune-related response criteria (iRECIST) | 5 years

OTHER OUTCOMES:
Health-related quality of life in all participants as assessed by EORTC Quality of Life Questionnaire Cancer QLC-C30 (Cancer 30-items). | 5 years
  All items are scored 1 (worse outcome) to 4 (better outcome) or 1 (worse outcome) to 7 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Change in circulating tumor DNA (ctDNA) levels after DOC1021 administration. | 5 years

IPD SHARING:
Plan to Share IPD: No